CLINICAL TRIAL: NCT00391846
Title: A Randomised, Single Blind, Multicentre, 9-month, Phase IV Study, Comparing Treatment Guided by Clinical Symptoms and Signs and NT-proBNP vs Treatment Guided by Clinical Symptoms and Signs Alone, in Patients With Heart Failure (HF) and Left Ventricular Systolic Dysfunction
Brief Title: Evaluation of Heart Failure Treatment Guided by N-terminal Pro B-type Natriuretic Peptide (NTproBNP) vs Clinical Symptoms and Signs Alone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2452L00010; EUDRACT No. 2006-001259-36; SIGNAL HF
Record Dates: First submitted 2006-10-19; First posted 2006-10-25 (Estimated); Results first posted 2012-06-18 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Heart Failure; Ventricular Dysfunction, Left
Keywords: Heart Failure; Ventricular Dysfunction; NTproBNP
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left; Ventricular Dysfunction | interventions — Captopril; Enalapril; Lisinopril; Ramipril; trandolapril; Bisoprolol; Carvedilol; Metoprolol; candesartan; candesartan cilexetil; Valsartan; Eplerenone; Spironolactone; Diuretics; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided by NT-proBNP (Other): Treatment guided by clinical symptoms and signs + NTproBNP
  Interventions: Drug: Captopril; Drug: Enalapril; Drug: Lisinopril; Drug: Ramipril; Drug: Trandolapril; Drug: Bisoprolol; Drug: Carvedilol; Drug: Metoprolol succinate; Drug: Candesartan; Drug: Valsartan; Drug: Eplerenone; Drug: Spironolactone; Drug: Diuretics; Drug: HF treatment according to Swedish guidelines; Procedure: Blood samples; Procedure: The Kansas City Cardiomyopathy Questionnaire (KCCQ)
- Not Guided by NT-proBNP (Other): Treatment guided by clinical symptoms and signs
  Interventions: Drug: Captopril; Drug: Enalapril; Drug: Lisinopril; Drug: Ramipril; Drug: Trandolapril; Drug: Bisoprolol; Drug: Carvedilol; Drug: Metoprolol succinate; Drug: Candesartan; Drug: Valsartan; Drug: Eplerenone; Drug: Spironolactone; Drug: Diuretics; Drug: HF treatment according to Swedish guidelines; Procedure: Blood samples; Procedure: The Kansas City Cardiomyopathy Questionnaire (KCCQ)

INTERVENTIONS:
Drug: Captopril
Drug: Enalapril
Drug: Lisinopril
Drug: Ramipril
Drug: Trandolapril
Drug: Bisoprolol
Drug: Carvedilol
Drug: Metoprolol succinate
Drug: Candesartan
  Other Names: Atacand
Drug: Valsartan
Drug: Eplerenone
Drug: Spironolactone
Drug: Diuretics
Drug: HF treatment according to Swedish guidelines
Procedure: Blood samples
Procedure: The Kansas City Cardiomyopathy Questionnaire (KCCQ)

SUMMARY:
The purpose is to study if HF treatment guided by NTproBNP in addition to clinical symptoms and signs is more effective than treatment guided by clinical symptoms and signs alone in patients with HF and left ventricular systolic dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Female/male, over 18 years with previously verified HF with left ventricular systolic dysfunction.
* New York Heart Association(NYHA) class II-IV,
* NTproBNP males>800 ng/L, females >1000 ng/L

Exclusion Criteria:

* Planned CV hospitalisation, stroke or acute myocardial infarction (MI) last 3 months,
* Mitral/aortic stenosis,
* Patients already receiving optimal HF treatment,
* Severe reduction of kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2006-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Sweden Medical Director, MD, Study Director — AstraZeneca; Hans Persson, MD, PhD, Principal Investigator — Danderyd Hospital, Sweden; Bjorn Eriksson, MD, Study Director — AstraZeneca
Locations (39):
- Sweden (39):
  - Research Site, Alvesta
  - Research Site, Arvika
  - Research Site, Bjuv
  - Research Site, Borensberg
  - Research Site, Bromma
  - Research Site, Dalby
  - Research Site, Eskilstuna
  - Research Site, Gagnef
  - Research Site, Gothenburg
  - Research Site, Hisings Kärra
  - Research Site, Huddinge
  - Research Site, Huskvarna
  - Research Site, Jönköping
  - Research Site, Kalmar
  - Research Site, Kungälv
  - Research Site, Lerum
  - Research Site, Lessebo
  - Research Site, Lidköping
  - Research Site, Lilla Edet
  - Research Site, Linköping
  - Research Site, Ludvika
  - Research Site, Lyckeby
  - Research Site, Malmo
  - Research Site, Moheda
  - Research Site, Motala
  - Research Site, Örebro
  - Research Site, Östersund
  - Research Site, Skanör
  - Research Site, Söderåkra
  - Research Site, Stenungsund
  - Research Site, Stocksund
  - Research Site, Timrå
  - Research Site, Uddevalla
  - Research Site, Ulricehamn
  - Research Site, Umeå
  - Research Site, Uppsala
  - Research Site, Vaxjo
  - Research Site, Västerås
  - Research Site, Västervik

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, parallel group, single blind, multicentre, 9-month study in chronic heart failure in patients with New York Heart Association classification of heart failure (NYHA) class II-IV, left ventricular systolic dysfunction and elevated NT-proBNP levels in the primary care setting.
Pre-assignment Details: At visit 1 was the NT-proBNP value measured at this value should be above 800 (females) or 1000 (males) before randomisation at visit 2. One patient from each group are excluded from the full analysis set (FAS) due to "total unavailability of efficacy data after randomisation".
Groups:
- Guided by NT-proBNP: Chronic heart failure treatment guided by clinical symptoms, signs and NT-proBNP
- Not Guided by NT-proBNP: Chronic heart failure treatment guided by clinical symptoms and signs
Period: Overall Study
Arm/Group | Guided by NT-proBNP | Not Guided by NT-proBNP
Started | 127 (Of the 127 randomised patients 8 were discontinued) | 125 (Of th 125 randomised patients 7 were discontinued)
Completed | 119 (119 completed patients includes 4 CV related deaths) | 118 (118 completed patients includes 5 CV related deaths)
Not Completed | 8 | 7
Not completed — Adverse Event | 4 | 1
Not completed — Did not meet the required elig. crit | 2 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Developed study specific DC criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guided by NT-proBNP | Not Guided by NT-proBNP | Total
Number analyzed (Participants) | 127 | 125 | 252
Age Continuous [Mean (Full Range); unit: Years] | 78 [57 to 92] | 77 [51 to 94] | 77 [51 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 42 | 72
  Male | 97 | 83 | 180
Electrocardiogram (ECG), Abnormal/Normal [Number; unit: Participants]
  Abnormal ECG | 115 | 113 | 228
  Normal ECG | 12 | 12 | 24
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 73 (11) | 75 (12) | 74 (11)
Pulse [Mean (Standard Deviation); unit: Beats/minute] | 71 (14) | 72 (14) | 72 (14)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 133 (21) | 135 (22) | 134 (21)

OUTCOME MEASURES:

1. Primary Outcome: Composite Value of 3 Variables After 9 Months: Cardiovascular Death (Days Alive), Cardiovascular Hospitalization (Days Out of Hospital), Heart Failure Symptoms (Symptom Score Subset of the Kansas City Cardiomyopathy Questionnaire - Questions 3,5,7,9)
Description: The non-parametric scale is constructed from 3 variables, modified after Cleland. Each patient receives a rank score from 1 to 246 (246-number of patients in the study). The lowest score receive patients who die (due to CV event), next patients still alive at end-of-study with the worst composite score, the best alive patients with 0 days in hospital and the largest improvement in the KCCQ (self-administered by patient symptom score, where the higher score reflect better health status). Scores will be summarized using non-parametric calculations. The mean of non-parametric scores is presented
Time Frame: 9 months
Population: In the above analysis regarding The number of participants analyzed the 'last observation carried forward' principle is used, as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Guided by NT-proBNP | Not Guided by NT-proBNP
Number analyzed (Participants) | 123 | 123
Scores on a scale | 118.6 (558) | 128.4 (558)

2. Secondary Outcome: Number of CV Deaths
Description: Number of deaths
Time Frame: 9 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Guided by NT-proBNP | Not Guided by NT-proBNP
Number analyzed (Participants) | 123 | 123
Participants | 4 | 5

3. Secondary Outcome: Number of Days in Hospital for CV Reason
Description: Each overnight stay is counted as one day. The lower the better
Time Frame: 9 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days in hospital
Arm/Group | Guided by NT-proBNP | Not Guided by NT-proBNP
Number analyzed (Participants) | 123 | 123
Days in hospital | 5.79 (6.63) | 5.94 (6.32)

4. Secondary Outcome: Changes in Heart Failure Symptoms
Description: Changes from baseline in the symptom score subset (question 3, 5, 7 and 9) of KCCQ (swelling, fatigue, shortness of breath, shortness of breath night time). KCCQ is a self-administered by patient symptom score, where higher score reflect better health status. Scale scores are transformed to a 0 to 100 range by subtracting the lowest possible scale score, dividing by the range of the scale and multiplying by 100. This mean that the KCCQ scale is from 0 to 100 with the higher value showing a better health status.
Time Frame: 9 months and baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Categorial scale
Arm/Group | Guided by NT-proBNP | Not Guided by NT-proBNP
Number analyzed (Participants) | 123 | 123
Categorial scale | 3.67 (20.02) | 6.11 (21.00)

5. Secondary Outcome: Changes in NT-proBNP Values Over Time in All Patients
Description: The 95% confidential interval (CI) is given as measure of dispersion
Time Frame: 9 months and baseline
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/L
Arm/Group | Guided by NT-proBNP | Not Guided by NT-proBNP
Number analyzed (Participants) | 123 | 123
ng/L | 2332.1 [1986.1 to 2738.4] | 2063 [1743.2 to 2442.7]

6. Secondary Outcome: Changes in Health-related Quality of Life
Description: Change range -100 to 100. The higher the better.
Time Frame: 9 months and baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: KCCQ overall score
Arm/Group | Guided by NT-proBNP | Not Guided by NT-proBNP
Number analyzed (Participants) | 123 | 123
KCCQ overall score | 1.739 (1.39) | 3.172 (1.39)

7. Secondary Outcome: Total Number of Titration Steps in Prescribed Heart Failure Treatment
Description: Each titration step in prescribed medication is counted as one step, either up or down. One step up indicates an increase of dose in prescribed medication and one step down indicates a decrease of dose in prescribed medication. The sum of steps is given as a score. Score is given for each arm as a total number of titration steps for all patients in arm.
Time Frame: 9 months
Population: as for outcome 1
Measure: Number; unit: Titration steps
Arm/Group | Guided by NT-proBNP | Not Guided by NT-proBNP
Number analyzed (Participants) | 123 | 123
Titration steps | 517 | 485

8. Secondary Outcome: Discontinuations
Description: Number of patients discontinued due to adverse events'
Time Frame: 9 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Guided by NT-proBNP | Not Guided by NT-proBNP
Number analyzed (Participants) | 127 | 125
Participants | 8 | 6

ADVERSE EVENTS:
Description: Only Serious Adverse Event were to be reported. Other Adverse Events (Non-Serious Adverse Events) were to be reported by investigators directly to MPA (Medical Product Agency) in accordance to local legislation.
Arm/Group | Guided by NT-proBNP | Not Guided by NT-proBNP
Serious Adverse Events (participants affected / at risk) | 46/127 | 41/125
Other Adverse Events (participants affected / at risk) | 0/127 | 0/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guided by NT-proBNP (N=127) | Not Guided by NT-proBNP (N=125)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Angina Pectoris (Cardiac disorders) | 2 | 1
Angina Unstable (Cardiac disorders) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 2
Aortic Stenosis (Vascular disorders) | 1 | 0
Artial Fibrillation (Cardiac disorders) | 2 | 3
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1
B-Cell Lymphoma (Blood and lymphatic system disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bleeding Varicose Vein (Vascular disorders) | 1 | 0
Blood Electrolytes Abnormal (Injury, poisoning and procedural complications) | 1 | 0
Blood Pressure Decreased (Injury, poisoning and procedural complications) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 2
Calculus Ureathral (Renal and urinary disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 12 | 7
Carotid Artery Stenosis (Vascular disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 2
Chest Pain (General disorders) | 0 | 2
Chronic Lymphocytic Leukaemia (Blood and lymphatic system disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 0
Death (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Diverticulitis (Infections and infestations) | 1 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Endocarditis (Infections and infestations) | 1 | 0
Fatigue (General disorders) | 0 | 1
Femur Fracture (General disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Tract Adenoma (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Headache (General disorders) | 0 | 1
Heamorrhage (Vascular disorders) | 0 | 1
Hepatic Failure (Renal and urinary disorders) | 1 | 0
Hip Fracture (General disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypertension (Vascular disorders) | 0 | 1
Intermittent Claudication (Vascular disorders) | 0 | 0
Intervertebral Disc Compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 1 | 0
Muscular Weakness (General disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 5 | 6
Odema Peripheral (General disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Peripheral Embolism (Vascular disorders) | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 4
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Pulmonary Odema (General disorders) | 1 | 0
Pyelonephritis (Renal and urinary disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 2
Respiratory Tract Infection Viral (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rib Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Right Ventricular Failure (Cardiac disorders) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 1
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Urosepis (Infections and infestations) | 0 | 1
Venous Thrombosis Limb (Vascular disorders) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 2 | 1
Vertigo (General disorders) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other